CLINICAL TRIAL: NCT01632592
Title: Abdominal Obesity, Cardiovascular Inflammation, and Effects of a Growth Hormone Releasing Hormone Analogue to Reduce Inflammation
Brief Title: Abdominal Obesity, Cardiovascular Inflammation, and Effects of Growth Hormone Releasing Hormone Analogue
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No funding available
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Steven K. Grinspoon, MD, Professor of Medicine, Harvard Medical School, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2012p-000917
Record Dates: First submitted 2012-06-27; First posted 2012-07-03 (Estimated); Last update posted 2014-01-24 (Estimated); Status verified 2014-01

CONDITIONS: Abdominal Obesity
MeSH Terms: conditions — Obesity, Abdominal | interventions — tesamorelin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Growth Hormone Releasing Hormone (Experimental): Growth Hormone Releasing Hormone analogue, 2mg subcutaneously every day for 12 months.
  Interventions: Drug: Tesamorelin
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tesamorelin — The Growth Hormone Releasing Hormone analogue tesamorelin, 2mg subcutaneously daily by injection
  Arms: Growth Hormone Releasing Hormone
Drug: Placebo — placebo given by injection 2mg subcutaneously daily
  Arms: Placebo

SUMMARY:
Obesity is strongly associated with risk of cardiovascular disease (CVD). Data increasingly suggest that visceral adipose tissue (VAT) accumulation -- or increased abdominal fat -- is particularly deleterious to cardiovascular health, but further study is needed to test this idea. Increased abdominal fat may also be associated with lower secretion of a hormone called growth hormone (GH), which helps the body burn fat. The current study aims to carefully characterize relationships between abdominal fat and CVD. In addition, by using a medication called growth hormone releasing hormone, which is a strategy to reduce abdominal fat, the investigators will test the hypothesis that abdominal fat contributes uniquely to increased arterial inflammation.

In the first part of this study, the investigators will investigate both lean (healthy weight) individuals and individuals with increased abdominal fat. The investigators will study their body composition, cardiovascular risk measures, insulin sensitivity, and growth hormone dynamics, with the hypothesis that abdominal fat, independent of general obesity, will be strongly associated with arterial wall thickening and atherosclerotic inflammation. The investigators will assess arterial wall thickness, plaque morphology, and atherosclerotic inflammation, and the investigators will determine associations between these variables and regional fat accumulation, with particular attention to abdominal fat.

The second, treatment part of the study will be only for individuals with increased abdominal fat who are found to have low growth hormone secretion. In that part of the study, the investigators will test the effects of a growth hormone releasing hormone (GHRH) analogue to reduce abdominal fat and, consequently, reduce arterial inflammation. The investigators hypothesize that abdominal fat reduction, independent of changes in growth hormone, will reduce arterial inflammation and arterial wall thickness.

ELIGIBILITY:
Inclusion/Exclusion Criteria:

Inclusion Criteria for Lean Controls:

1. Men and women age 18-55y
2. BMI > 18.5 and < 25 kg/m2
3. Waist circumference < 102 cm in men and <88cm in women

Inclusion criteria for Abdominal Obesity:

1. Men and women age 18-55y
2. BMI ≥ 30kg/m2
3. Abdominal obesity as defined by waist circumference ≥ 102 cm in men and ≥ 88 cm in women
4. Relative GH deficiency as demonstrated by peak GH to arginine/GHRH stimulation test of < 9mcg/L (for treatment portion only)
5. Negative age-appropriate screening for cancer performed by primary care physician (e.g., negative mammogram if F > 50yo) (For treatment portion only)

Exclusion criteria for all subjects:

1. Obesity due to known secondary causes
2. Use of weight-lowering drugs or previous weight loss surgery
3. Use of gonadal steroids, GH, GHRH, glucocorticoids, megesterol acetate, antidiabetic agents, or any other hormonal medication judged by the investigator to be inappropriate within the past 6 months. Use of physiologic testosterone replacement will be allowed.
4. Statin use
5. Known coronary artery disease or peripheral vascular disease, or any history of stroke or significant chest pain
6. Known auto-immune or inflammatory disease
7. Any surgery or significant injury (including fracture or other trauma) within the past 6 months
8. Hemoglobin < 11g/dL, fasting glucose > 126mg/dL, creatinine <1.5mg/dL, or AST > 2.5x upper limit of normal
9. FSH > 20 IU/L (women only)
10. Positive urine pregnancy test, actively seeking pregnancy, or breastfeeding
11. Prior history of pituitary disease, pituitary surgery, or head irradiation, or any other condition known to affect pituitary function
12. Infectious illness in the past 3 months, or chronic infectious illness
13. Allergy to iodine containing contrast media
14. Active illicit drug use
15. For women of childbearing potential, failure to use an acceptable form of non-hormonal birth control
16. Active malignancy: For the treatment part of the study, all active malignancy will be excluded. For the observational part of the study (which involves no intervention) basal cell carcinoma and low grade cervical or anal intraepithelial neoplasms will be allowed.
17. History of colon cancer (treatment part only)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2014-01; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
aortic "target to background ratio" (Aortic TBR) | 12 months
  aortic target-to-background ratio is a measure of the inflammation in the wall of the aorta that is made by positron emission tomography (PET) scanning in conjunction with computed tomography (CT) scanning.

CONTACTS AND LOCATIONS:
Overall Officials: Steven Grinspoon, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States